CLINICAL TRIAL: NCT06694688
Title: Evaluation of the Contribution of Lower Limb and/or Abdominal Compression on Orthostatic Hypotension.
Acronym: HYPOFLEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gérond'if (Other)
Collaborators: Thuasne (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-A00027-40
Record Dates: First submitted 2024-11-08; First posted 2024-11-19 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Orthostatic Hypotension
Keywords: orthostatic hypotention; abdominal compression; Lower limb compression
MeSH Terms: conditions — Hypotension, Orthostatic

STUDY DESIGN:
Intervention Model Description: 44 patients will be included in this study. Randomization will be carried out to determine the order of the 5 conditions studied:
  * No compression,
  * Class 2 compression socks,
  * Class 3 compression socks,
  * Class 2 compression tights,
  * Dynabelt abdominal belt + Class 2 compression socks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- a single group of patients (Other): Subject will undergo the following 5 conditions in the cross-over scheme as determined by the randomization:
  No compression, Class 2 compression socks, Class 3 compression socks, Class 2 compression tights and Dynabelt abdominal belt + Class 2 compression socks
  .
  Interventions: Diagnostic Test: the supine/standing postural change test

INTERVENTIONS:
Diagnostic Test: the supine/standing postural change test — The prevalence of orthostatic hypotension will be characterized by the percentage of patients with a decrease of ≥ 20mmHg in systolic blood pressure or ≥ 10mmHg in diastolic blood pressure following the supine/standing postural change position.

SUMMARY:
Orthostatic hypotension (OH) is associated with an increased risk of myocardial infarction, stroke, heart failure and neurocognitive disorders. In the elderly, OH is an independent predictor of falls and mortality. Non-drug treatments are used as the first-line treatments. Among non-drug treatments, compression of the lower limbs and abdominal compression have been shown to help reduce OH and associated symptoms. As these studies were solely based on ankle-to-thigh bandages, the effectiveness of other medical devices developed, such as compression socks and tights, needs to be evaluated. In addition, data comparing the efficacy and tolerability of several approaches, single or combined, of several levels of compression, provided by socks, tights and an abdominal belt are scarce. The HYPOFLEX study aims to provide new data to enable better management of OH.

DETAILED DESCRIPTION:
Patients will be recruited from a single center, over a 12-month inclusion period. The clinical investigation will focus on CE-marked Class I medical devices, used for their intended purpose, as part of a post-market clinical follow-up with additional non-invasive, non-invasive procedures. Randomization will be carried out to determine the order of the 5 conditions studied:

* No compression,
* Class 2 compression socks,
* Class 3 compression socks,
* Class 2 compression tights,
* Dynabelt abdominal belt + Class 2 compression socks. Conditions will be tested over half a day.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 60 or over,
* Patients hospitalized at Broca Hospital with orthostatic hypotension,
* Patient able to stand,
* Patient who has been medically stable for at least 48 hours,
* Patient whose measurements are compatible with Thuasne compression device sizes,
* Patient having been informed, having received answers to his questions and having signed the informed consent form prior to his participation in the study,
* Patient affiliated or entitled to a social security number.

Exclusion Criteria:

* Patients presenting, according to the investigator, a contraindication to lower limb and/or abdominal compression,
* Patients presenting any contraindication mentioned in the instructions for use of the medical devices under investigation.
* Patient presenting, according to the investigator, a major cognitive impairment incompatible with participation in a clinical trial,
* Patient taking part in another clinical investigation conducted to establish the conformity of a medical device having an impact on the outcomes,
* Vulnerable patient according to article L1121-6 of the Public Health Code, subject to a judicial protection measure or incapable of consenting to a clinical trial or incapable of giving informed consent.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Compare the blood pressure reduction induced by supine/standing postural change in the absence and presence of lower limb compression. | 12 months
  Decrease in systolic BP when moving from the supine to the standing position, using a semi-automatic blood pressure monitor (Dynamap type):
  * supine BP: average of 3 measurements taken after a rest of at least 5 minutes
  * BP in upright position: lowest value of measurements obtained every minute for 5 minutes after rising, Without compression and with class 2 compression of the lower limbs.

SECONDARY OUTCOMES:
Decrease in systolic blood pressure when moving from the supine to the upright position | 12 months
  The following evaluation criteria will be compared in the absence and presence of compression and between the different compression devices:
  * The difference between supine SBP/DBP (average of last 3 measurements) and standing SBP/DBP (lowest value of 5 measurements) will be calculated,
  * The prevalence of orthostatic hypotension will be characterised by the percentage of patients with a decrease in systolic BP ≥ 20mmHg or ≥ 10mmHg in diastolic BP following the supine/standing postural change position,
  * The time to onset of orthostatic hypotension will be calculated from the 5 measurements of BP measured in orthostasis,
Severity of orthostatic hypotension | 12 months
  The severity of orthostatic hypotension will be assessed by the percentage of patients with an orthostatic systolic BP <90mmHg, following the supine/standing postural change position,
  - Symptoms associated with orthostatic hypotension will be assessed using the Orthostatic Hypotension Symptoms Assessment questionnaire (OHQ), consisting of 6 questions at the end of all pressure measurements.
Characterize orthostatic hypotension | 12 months
  Characterize orthostatic hypotension at inclusion (neurogenic, hypovolemic, cardiogenic, drug-induced).
Evaluate patient satisfaction and tolerance | 12 months
  Evaluate patient satisfaction and tolerance with the use of compression devices.

CONTACTS AND LOCATIONS:
Locations (1):
- Broca Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No